CLINICAL TRIAL: NCT02012114
Title: A Cohort of Patients With Cystinosis : Compliance to Cysteamine and Neurological Complications
Acronym: Crystobs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010-605
Record Dates: First submitted 2012-12-11; First posted 2013-12-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cystinosis
Keywords: Cystinosis, compliance, cysteamine, neurological assessments
MeSH Terms: conditions — Cystinosis; Patient Compliance | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cysteamine Bitartrate (No Intervention): Single arm study. Subjects receive their current oral form of cysteamine bitartrate treatment : Cystagon® or RP103
  Interventions: Other: Cysteamine bitartrate

INTERVENTIONS:
Other: Cysteamine bitartrate — No intervention

SUMMARY:
Preventing late onset of Cystinosis such as neurological complications and improving compliance to cysteamine treatment remain major challenges in management of subjects with cystinosis.

This study is designed to describe the relationship between compliance of patients with cystinosis treated with cysteamine and treatment efficacy and to understand the pathophysiologic mechanism of neurological disorders. Is cysteamine crossing the blood brain barrier? What is the impact of cystine accumulation in Cerebro Spinal Fluid and Central Nervous System? Our Primary objective is to study the relationship between compliance of patients treated with cysteamine and the WBC cystine level.

Secondary, the study will assess relationship between compliance to cysteamine and its neurological consequences.

The expected duration of the study is 48 months. The enrolment period is 24 months and the study participation of each subject is 24 months. Eligible participants are male and female (age > 4 years) with confirmed diagnosis of cystinosis and receiving any oral cysteamine treatment: Cystagon or RP103.

The compliance under cysteamine is measured using electronic devices, accountability of study treatment, and information in patients' diary. Specific memory and visuoperceptual tests are performed at the beginning and at the end of patients'participation. Nuclear Magnetic Resonance spectroscopy is used to detect possible sites of cystine accumulation in the CNS and their relationship with compliance to cysteamine treatment. NMRS is also used to establish a relationship with the neuropsychological status of the subject.

To describe absorption, distribution and elimination of cysteamine, and its metabolic pathways, and to determine the concentration effect and dose effect relationship, blood samples are performed at each study visit. A lumbar puncture is also proposed to participants to verify if cysteamine is crossing the blood brain barrier. New tools are used to compare metabonomic networks in patients with cystinosis and their controls.

ELIGIBILITY:
* Male and female subjects with confirmed diagnosis of nephropathic cystinosis (defined by clinical signs and WBC cystine level).
* Age > 4 years.
* Subjects receiving any oral cysteamine treatment: Cystagon or RP103.
* Sexually active female subjects of childbearing potential must agree to utilize the same acceptable form of contraception from day 1 through completion of the study.
* Subjects or their parent or legal guardian must provide written informed consent prior to participation in the study.
* Subjects covered by or having the right to social security.

Exclusion Criteria:

* Subjects with known hypersensitivity to cysteamine and penicillamine.
* Females who are nursing, planning a pregnancy, known or suspected to be pregnant, or with a positive urinary pregnancy test.
* Subjects who, in the opinion of the Investigator, are not able or willing to comply with the protocol.
* Contra-indication to MRI assessment

CONTROLS FOR METABONOMIC ASSESSMENTS

Inclusion Criteria:

- Age and sex matched to study population: Age range: patients aged 4 to 5 years, 6 to 11 years, patients aged 12 to 17 years, adult patients: 18 or above.

Sex: male or female

* Subjects or their parent or legal guardian must provide written informed consent prior to participation in the study.
* Subjects covered by or having the right to social security.

Exclusion Criteria:

- Any uropathology or nephropathology.

CONTROLS FOR NMRS ASSESSMENTS

Inclusion Criteria:

- Age and sex matched to study population: Age range: patients aged 4 to 5 years, 6 to 11 years, patients aged 12 to 17 years, adult patients: 18 or above.

Sex: male or female

* Subjects or their parent or legal guardian must provide written informed consent prior to participation in the study.
* Subjects covered by or having the right to social security.

Exclusion Criteria:

* Any uropathology or nephropathology.
* Any neurological and/or psychiatric disorder
* Contra-indication to MRI assessment.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12-05 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
WBC cystine levels | Day1and every three months : Month1, Month3, Month6, Month9, Month12, Month15, Month18, Month21 and Month24.
  PD measurements will be performed at D1, M1, M3, M6, M9, M12, M15, M18, M21 and M24.
  Compliance under cysteamine will be measured from D1 to M24 using electronic devices (date and time of bottle opening are recorded), accountability of study treatment and information of patients' diary. Compliance measurement between two consecutive study visits will be expressed as the proportion of the observed number of opening compared to the expected number and the cumulated dose taken compared to the expected dose.Compliance will be first considered as a dichotomous variable, the compliance being described as satisfactory if greater than 95% during a specific period.Compliance will then be considered as a quantitative variable

SECONDARY OUTCOMES:
Presence or absence and accountability of cystine crystals. | Every 6 month : Month1, Month6, Month12, Month18, Month24
  Eye examination
Memory and visuoperceptual tests repeated during the study | at Day 1 and two years
presence or absence of cystine accumulation, determination of the sites of cystine accumulation in the CNS and relationship with the compliance to cysteamine treatment, relationship with neuropsychological status. | at Month 1 and two years
  NMRS assessments
Concentration of cysteamine in the CSF, associated to a measurement of the CSF pressure | at any visit
concentration of cysteamine in blood (measured by toxicological HPLC analysis with fluorescence detection) | at Day1 and every 3 months : month1, month3, month6, month9, month12, month15, month18, month21, month24
discrimination of urine and blood samples,from metabolic spectroscopic data obtained by nuclear magnetic resonance. | Every 3 months during 6 months and every 6 months to month 6 until two years
  Perturbed metabolic network resulting from the intake of cysteamine in comparison to controls,using urine and blood samples available for patients with cystinosis and their controls
Concentration effect, dose effect model. | at month 6
  pharmacokinetic profile and 2 timepoints pharmacodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Cochat Pierre, PUPH, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Gaillard S, Roche L, Lemoine S, Deschenes G, Morin D, Vianey-Saban C, Acquaviva-Bourdain C, Ranchin B, Bacchetta J, Kassai B, Nony P, Bodenan E, Laudy V, Rouges C, Zarrabian S, Subtil F, Mercier C, Cochat P, Bertholet-Thomas A. Adherence to cysteamine in nephropathic cystinosis: A unique electronic monitoring experience for a better understanding. A prospective cohort study: CrYSTobs. Pediatr Nephrol. 2021 Mar;36(3):581-589. doi: 10.1007/s00467-020-04722-0. Epub 2020 Sep 9. PMID 32901297